CLINICAL TRIAL: NCT03925116
Title: Impact of a Contraceptive Pathway on Contraception Continuation Rates
Brief Title: Contraceptive Pathway and Contraception Continuation Rates
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: budget
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Adrian C Balica, MD, Associate Professor, Dept. Ob/Gyn, RWJMS, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro2018002901
Record Dates: First submitted 2019-03-26; First posted 2019-04-23 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Contraceptive Usage
Keywords: contraceptive pathway; continuation
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Intervention Model Description: randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual care (No Intervention): women who present for birth control to the gynecology office will see their physician in the usual fashion for review, counseling and contraception decision/initiation.
  Follow up phone call will be done at 2 weeks, 3, 6 and 12 months to discuss contraception initiation and continuation.
- Contraceptive pathway (Experimental): Women who present for birth control to the gynecology office will be recognized by the front desk and offered a tablet which which will:
  1. collect relevant medical history
  2. provide educational material on birth control options
  3. provide a link to bedsider.com for further information
  They will then discuss the tablet information/history with the medical assistant, who will answer any remaining questions. They will then see the physician/APN.
  Follow up phone call will be done at 2 weeks, 3, 6 and 12 months to discuss contraception initiation and continuation.
  Interventions: Other: COntraceptive pathway

INTERVENTIONS:
Other: COntraceptive pathway — alternative way of aiding patients in deciding contraception method
  Arms: Contraceptive pathway

SUMMARY:
Women seeking contraception will be randomized to "usual care" or to a "Contraceptive Pathway"

DETAILED DESCRIPTION:
Patients who present to the gynecology clinic for an annual, postpartum or contraceptive visit will be asked if they are interested in obtaining contraception by the front desk staff. If they respond yes, they will be seen in a triage or exam room by study personnel/medical assistant (MA) who will ask them if they would like to participate in the study, review the study and then randomize them to either the contraceptive pathway or usual care. The randomization will be done by opening sequentially numbered envelopes once they consent and while in the triage/exam room.

Patients triaged to the pathway will be handed an electronic tablet questionnaire while they are waiting to see the physician/(Advanced practice nurse (APN). The tablet contains a link to bedside.org, a public website which reviews contraceptive options. Vital signs will be collected as per usual care and recorded on both the questionnaire and in the electronic medical record(EMR). Study personnel will be available to offer the patient additional information on their choice of contraception or assist them with the link for information. The completed survey will be printed and placed in the subject room for review by the physician/APN. A copy will be kept in the subject binder and another will be scanned into the EMR.

Patients triaged to usual care will wait for their physician without the pathway questionnaire and will be asked the usual questions by the MA which will be recorded in the EMR. Vital signs will be collected and recorded in the EMR.

The physician/APN will see the subject as usual, review either the questionnaire or the EMR, review contraception options and initiate the contraception.

At completion of the visit, all woman will be asked if she would complete a satisfaction survey for her visit. She will be called at 2 weeks, 3, 6 and 12 months to discuss contraception initiation and continuation.

ELIGIBILITY:
Inclusion Criteria

* Women at risk for pregnancy
* Women able to read and write in English

Exclusion Criteria

* Women who have undergone permanent sterilization
* Women not sexually active with a male partner
* Women who intend to become pregnant in the next 12 months

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-01-03 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Continued Use of Contraception at 1 year | 1 year
  The difference in contraception continuation rates will be compared between the Contraceptive Pathway group and the Usual care group, based on follow up phone calls at 3 weeks, 6 months and 1 year

SECONDARY OUTCOMES:
Subject satisfaction with contraceptive counseling | at initial office visit/immediate
  Subjects will complete a Likert scale 1 - 5 with 1 being most and 5 being least satisfied with the contraceptive counseling. Responses will be compared between the Contraceptive Pathway and Usual care group
Pregnancy rates | 1 year
  At each phone call, interval pregnancy rates will be collected and compared between subjects in the Contraceptive pathway vs usual care

CONTACTS AND LOCATIONS:
Overall Officials: Adrian C Balica, MD, Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (1):
- Clinical Academic Building. 125 Paterson Street, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: public website with contraceptive information — http://bedsider.com